CLINICAL TRIAL: NCT03673319
Title: The Influence of Patient Expectation in Dry Needling Induced Analgesia
Brief Title: The Patient Expectation in Dry Needling and Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI18/087
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive expectative (Experimental): Participants in the positive expectation group will be told that DN procedure: "is a very effective form of treatment used to treat neck-shoulder pain and it is expected to reduce your perception of pressure pain"
  Interventions: Procedure: Dry needling with positives expectation
- Neutral expectatives (Experimental): Participants in the neutral expectation group will be told that DN procedure: "is a form of treatment used to treat neck-shoulder pain that has unknown effects on your perception of pressure pain"
  Interventions: Procedure: Dry needling with neutral expectation

INTERVENTIONS:
Procedure: Dry needling with positives expectation — DN procedure: "is a very effective form of treatment used to treat neck-shoulder pain and it is expected to reduce your perception of pressure pain"
  Arms: Positive expectative
Procedure: Dry needling with neutral expectation — DN procedure: "is a form of treatment used to treat neck-shoulder pain that has unknown effects on your perception of pressure pain"
  Arms: Neutral expectatives

SUMMARY:
This study will evaluate placebo mechanisms related to dry needling(DN) trying to determinate whether an additive effect occurs when DN is provided with an instructional set known to enhance placebo analgesia. External manipulation of patient expectation for receiving DN will be performed, in a similar way as has been already done in studies investigating the influence of expectation on spinal manipulative therapy interventions. The main purpose of this study will be therefore to determine, for the first time, how subjects' expectation about the effect of DN influences the resultant hypoalgesia. Analgesic effects of DN will be assessed using the conditioned pain modulation (CPM) paradigm, which has not been previously evaluated in relation to DN.

DETAILED DESCRIPTION:
Just before DN intervention, participants will receive a positive or a neutral expectation instructional set regarding effects of a DN technique on pain perception. This instructional set will be randomly allocated to each patient.

Participants in the positive expectation group will be told that DN procedure: "is a very effective form of treatment used to treat neck-shoulder pain and it is expected to reduce your perception of pressure pain". Participants in the neutral expectation group will be told that DN procedure: "is a form of treatment used to treat neck-shoulder pain that has unknown effects on your perception of pressure pain".

DN intervention An experienced and trained physical therapist will provide DN to all the subjects. This researcher will be blinded to the specific expectation instructional set the participant receives. Participants will receive one session of DN treatment for the active Myofascial Trigger Points(MTrP) located at the upper trapezius muscle. They will be placed in a prone position on the examination table. Solid filament needles of 0.30 mm diameter and 40 mm length will be used. The needle will be inserted into the skin over the palpated MTrP using pincer palpation, and slowly advanced perpendicularly until it reaches the MTrP and a twitch response is elicited.

ELIGIBILITY:
Inclusion Criteria:

* neck pain (≥3 months of duration)
* VAS of 4-5 of pain.
* Presence of at least one active MTrP located at the upper trapezius.

Exclusion Criteria:

* Patients with previous cervical spine or shoulder surgery.
* Cervical spine radiculopathy or myelopathy.
* Systemic disease.
* Fibromyalgia.
* Pregnancy.
* Using sedative drugs.
* Needle phobia.
* Bleeding disorder.
* anticoagulant medication.
* Previous experience with DN for myofascial pain.
* Skin lesion and infection or inflammatory oedema at the MTrPs site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity: Visual Analog Scale (VAS) | Change from Baseline at after intervention
  The investigators use a Visual Analog Scale (VAS) to determine the intensity of the patient's current pain before, during DN and immediately after DN. We will follow the paradigm of Conditioned pain modulation (CPM) paradigm. CPM will be induced by inflating an occlusion cuff (conditioning stimulus) at the arm, at the opposite side from the affected upper trapezius.The VAS is a 100-mm line, oriented horizontally, with one end representing "no pain"(the best value) and the other end representing "worst pain" (the worse value). Subjects will be asked to rate their current pain with a mark on the scale.

SECONDARY OUTCOMES:
Pain Pressure Threshold (PPT) | Change up 1 hour
  The PPT serves to determine the sensitivity of hiperalgesic focus. The investigators will done it with one algometer.
  Lower values are a worse result. Higher values are a better result.
Dry needling pain | Change up 1 hour
  The investigators use a Visual Analog Scale (VAS) to determine the intensity of the patient's pain during DN intervention.The VAS is a 100-mm line, oriented horizontally, with one end representing "no pain" (the best value) and the other end representing "worst pain" (the worse value). Subjects will be asked to rate their current dry needling pain with a mark on the scale.
Dry needling anxiety | Change up 1 hour
  The investigators use a Visual Analog Scale (VAS) to determine the anxiety of the patient during DN.The VAS is a 100-mm line, oriented horizontally, with one end representing "no anxiety"(the best value) and the other end representing "worst anxiety"(the worse value). Subjects were asked to rate their current dry needling anxiety with a mark on the scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, Phd, Principal Investigator — Alcala University
Locations (2):
- Spain (2):
  - Institut Physiotherapy AND pain, Alcalá de Henares, Madrid
  - Grupo Fisioterapia y Dolor, Alcalá de Henares, Madrid

IPD SHARING:
Plan to Share IPD: No
The IDP does not exist